Feasibility and Safety Study PI: Baburao Koneru, MD, MPH



Department of Surgery/Division of Liver Transplant and Hepatobiliary Surgery Rutgers, The State University of New Jersey 185 South Orange Avenue, Medical Science Building G595 Newark, NJ 07103

p. 973-972-9599 f. 973-972-9292

#### I. SUBJECT CONSENT TO TAKE PART IN A RESEARCH STUDY

**TITLE OF STUDY:** Remote Ischemic Conditioning (RIC) in Recipients of Brain Death Donor Livers – A Feasibility and Safety Study

### Principal Investigator: Baburao Koneru, MD, MPH

This consent form is part of an informed consent process for a research study and it will provide information that will help you to decide whether you wish to volunteer for this research study. It will help you to understand what the study is about and what will happen in the course of the study.

If you have questions at any time during the research study, you should feel free to ask them and should expect to be given answers that you completely understand.

After all of your questions have been answered, if you still wish to take part in the study, you will be asked to sign this informed consent form.

You are not giving up any of your legal rights by volunteering for this research study or by signing this consent form.

Who is conducting this research study?

Dr. Baburao Koneru, MD, MPH is the Principal Investigator of this research study. A Principal Investigator has the overall responsibility for the conduct of the study. However, there are often other individuals who are part of the research team.

Dr. Koneru may be reached at (973) 972-9599; His office address is Room G-595, 185 South Orange Avenue, Newark, NJ 07101

The study doctor, Dr. Koneru, or another member of the study team will also be asked to sign this informed consent. You will be given a copy of the signed consent form to keep.

Who might benefit financially from this research?

Research studies like this one are designed to determine whether a particular treatment is safe and effective. In certain research studies conducted at Rutgers University, a party or parties (Rutgers University, the investigatory or a drug company) may gain financial benefits.

However, in this particular research study, there are no financial benefits to anyone.

Why is this study being done?

Several complications may happen after a liver transplant operation. Breathing problems may require you to be on a machine more than a day or two. Kidneys may make less urine than what is needed. Livers suffer damage when transplanted from one person to another. This damage could further increase complications after the transplant. The study doctors are interested in

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

decreasing complications after liver transplants. They are doing research with a simple treatment called CONDITIONING. This is not a medicine. In CONDITIONING rubber cuffs (similar to those used to check blood pressure) are put on the thigh. They are filled with air for 5 minutes and then air is let out for another five minutes. This is repeated 3 times.

Other doctors have found that patients getting this type of CONDITIONING do better after heart operations. Their kidneys work better. This study's doctors want to make sure CONDITIONING is safe in patients receiving liver transplants and CONDITIONING does not cause excessive amounts of pain when done after surgery. Also, this study's doctors want to see if CONDITIONING would improve your breathing, and make your kidneys and liver work better after transplant.

Why have you been asked to take part in this study?

You are about to receive a liver transplant. Therefore, we are asking that you consider participation in this study.

### Who may take part in this study? And who may not?

You are eligible to participate in this study if

1) You agreed to receive a liver transplant

- 2) You are either on or about to be put on the waiting list for a liver transplant
- 3) You are 18 years of age or older
- 4) You sign a research consent form
- 5) You may have diabetes, but take only insulin or metformin for sugar control
- 6) You do not have any serious circulation or nerve problems in your legs

You are not eligible to participate in this study if you

- 1) Have amputations in one or both legs
- 2) Have diabetes and take certain tablets for sugar control
- 3) Have circulation and nerve problems in your legs
- 4) Take nitrate pills for heart or other medical problems
- 5) Are extremely overweight
- 6) Are pregnant

How long will the study take and how many subjects will participate?

You will take part in this study for 90 days after your transplant. Once you are discharged, no extra trips to the hospital are needed for the research. Approximately thirty patients like you will participate in this study.

What will you be asked to do if you take part in this research study?

As part of this study, you will receive CONDITIONING treatments a total of 6 times during and after your liver transplant.

During your transplant, a rubber cuff will be placed on your thigh. The rubber cuff will be pumped with air for 5 minutes. Then the air will be let out and left for 5 minutes. This will be repeated for a total of 3 times. This constitutes one CONDITIONING treatment. The same treatment will be repeated again at the end of your operation before you leave the operating room. After the transplant, the same thing will be done once daily in the morning for 4 days.

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

What are the risks and/or discomforts you might experience if you take part in this study?

1) When study doctors do CONDITIONING during transplant you will not know and feel anything. Depending on your medical condition you may be fully awake by the time study doctors do CONDITIONING after the transplant. If you are awake, you may feel some discomfort or slight pain in the leg for a minute or two when the rubber cuff is pumped with air. Also, you will experience some tingling and "pins and needles" for a minute or two when the air is let out. The goal of this study is to make sure this pain is not excessive and that CONDITIONING does not interfere with the care you otherwise receive.

If you have significant pain from the conditioning, you have the right to opt out of receiving further conditioning. If you do so, the study doctors will still use information about you. You may also withdraw your consent for the use of your data, but you must do this in writing to Baburao Koneru, M.D, MPH, MSB G-599, 185 South Orange Avenue, Newark NJ 07101.

Are there any benefits for you if you choose to take part in this research study? You may have fewer complications from liver transplantation. If conditioning makes your lungs work better, you may get off the breathing machine sooner. If conditioning makes your lungs, kidneys and liver work better, you may leave the ICU and the hospital sooner.

However, it is possible that you might receive no direct personal benefit from taking part in this study.

What are your alternatives if you don't want to take part in this study? The alternative is to proceed with the liver transplant without participating in this study.

How will you know if new information is learned that may affect whether you are willing to stay in this research study?

During the course of the study, you will be updated about any new information that may affect whether you are willing to continue taking part in the study. If new information is learned that may affect you after the study or your follow-up is completed, you will be contacted.

Will there be any cost to you to take part in this study?

Your participation in this study will be free of cost to you. You or your insurance carrier will be billed for your routine care.

Will you be paid to take part in this study?

You will not be paid for your participation in this research study.

How will information about you be kept private or confidential?

All efforts will be made to keep your personal information in your research record confidential, but total confidentiality cannot be guaranteed. Information collected about you will be in paper records and in a computer dedicated to research use. The paper records will be stored in locked file cabinets in locked rooms. Access to computers containing information about you will be restricted by passwords. Also, those computers will be stored in locked rooms. Only people connected directly with the study will see or receive information about you.

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

A description of this clinical trial will be available on ClinicalTrials.gov, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

What will happen if you are injured during this study?

Subjects in this study will be exposed to certain risks of personal injury in addition to those associated with standard forms of treatment, which include the risks associated with having a liver transplant. Your regular doctors and nurses have already provided you with that information in your meetings with them and via the Transplant Handbook.

In addition, it is possible that during the course of this study, new adverse effects of CONDITIONING that result in physical injury may be discovered. The University will make appropriate referrals for medical and/or dental treatment for subjects who sustain personal injuries or illnesses as a direct consequence of participation in the research. The subject's health insurance carrier or other third-party payer will be billed for the cost of this treatment; provided that the University shall not submit to federally funded programs, e.g., Medicare, Medicaid or CHAMPUS, for reimbursement first if submission to such programs is prohibited by law. The University will provide no financial compensation. No other type of assistance is available from the University.

What will happen if you do not wish to take part in the study or if you later decide not to stay in the study?

Participation in this study is voluntary. You may choose not to participate or you may change your mind at any time.

If you do not want to enter the study or decide to stop participating, your relationship with the transplant team will not change, and you may do so without penalty and without loss of benefits to which you are otherwise entitled.

You may also withdraw your consent for the use of your data, but you must do this in writing to Baburao Koneru, M.D, MPH, MSB G-599, 185 South Orange Avenue, Newark NJ 07101. At any time, the study doctor can take you out of this study because it would not be in your best interest to stay in it. Your study doctor can stop treatment even if you are willing to stay in the study.

Who can you call if you have any questions?

If you have any questions about taking part in this study or if you feel you may have suffered a research related injury, you can call the study doctor:

> Baburao Koneru, MD, MPH Department of Surgery 973-972-9599

If you have any questions about your rights as a research subject, you can call:

IRB Director, Newark (973)-972-3608

And

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

> Human Subjects Protection Program, Newark (973) 972-1149

What are your rights if you decide to take part in this research study?

You have the right to ask questions about any part of the study at any time. You should not sign this form unless you have had a chance to ask questions and have been given answers to all of your questions.

### PERMISSION (Authorization) TO USE OR SHARE HEALTH INFORMATION THAT **IDENTIFIES YOU FOR A RESEARCH STUDY**

Information about you and your health is personal and private, so this information generally cannot be used in research without your written permission. The next few paragraphs tell you about how researchers want to use and share your health information in this research study. Your information will only be used as described here or as allowed or required by law. Ask questions if you do not understand any part of the research or the use of your health information. If you sign this consent form, you agree to let the researchers use your information in the research and share it with others as described below.

What is the purpose of the research and how will my information be used?

You are being invited to take part in this research study, which is described at the beginning of this form. The purpose of collecting and using your health information for this study is to help researchers answer the questions that are being asked in the research.

### What information about me will be used?

- All information in your medical record except for dental records and financial and billing information.
- Medical information regarding your donor.

Who may use, share or receive my information?

The research team may use or share your information collected or created for this study with the following people and institutions:

- Rutgers University researchers involved in the study;
- The Rutgers University Institutional Review Board and Compliance Boards;
- The Office for Human Research Protections in the U.S. Dept. of Health and Human Services.

Those persons or organizations that receive your information may not be required by Federal privacy laws to protect it and may share your information with others without your permission, if permitted by the laws governing them.

Will I be able to review my research record while the research is ongoing? No. We are not able to share information in the research records with you until the study is over. To ask for this information, please contact the Principal Investigator, the person in charge of this research study.

Do I have to give my permission?

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

No. You do not have to permit use of your information. But, if you do not give permission, you cannot take part in this research study. (Saying no does not stop you from getting medical care or other benefits you are eligible for outside of this study.)

If I say yes now, can I change my mind and take away my permission later?

Yes. You may change your mind and not allow the continued use of your information (and to stop taking part in the study) at any time. If you take away permission, your information will no longer be used or shared in the study, but we will not be able to take back information that has already been used or shared with others. If you say yes now but change your mind later for use of your information in the research, you must write to Baburao Koneru, MD, MPH, Room G-595, 185 South Orange Avenue, Newark, NJ 07101, and tell him of your decision.

How long will my permission last?

Your permission for the use and sharing of your health information will last until the end of the research study.

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

| AGREEMENT TO PARTICIPATE | |
|---|---|
| 1. Subject consent: | |
| I have read this entire form, or it has been read to me, and I believe that I understand been discussed. All of my questions about this form or this study have been answere | what has |
| Subject Name: | ···· |
| Subject Signature:Date: | |
| 2. Signature of Investigator/Individual Obtaining Consent: | |
| To the best of my ability, I have explained and discussed the full contents of the studincluding all of the information contained in this consent form. All questions of the subject and those of his/her parent or legally authorized representative have been ac answered. | research |
| Investigator/Person Obtaining Consent (printed name): | |
| Signature:Date: | |
| 3. Signature of Consent Process Witness: I have observed the consent process, which included a description of the purposes a procedures of this Study and an opportunity for questions and answers about this St attest that I am not the subject, his/her guardian or authorized representative, or a re on this study and can attest that the requirements for informed consent to the medic have been satisfied. | and<br>tudy. I<br>esearcher |
| Signature of Witness Printed Name of Witness Date | |

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH



Department of Surgery/Division of Liver Transplant and Hepatobiliary Surgery Rutgers, The State University of New Jersey 185 South Orange Avenue, Medical Science Building G595 Newark, NJ 07103

p. 973-972-9599 f. 973-972-9292

### II. SURROGATE CONSENT TO TAKE PART IN A RESEARCH STUDY

TITLE OF STUDY: Remote Ischemic Conditioning (RIC) in Recipients of Brain Death Donor Livers – A Feasibility and Safety Study

### Principal Investigator: Baburao Koneru, MD, MPH

Under certain circumstances, an individual can give consent for another person to take part as a Subject in this Research Study (hereinafter "Study") because the Subject is unable to consent to this Study and the Subject has not expressed opposition either to this Study or to the determination of incapacity. This individual is called the Legally Authorized Representative, or Surrogate, and is providing Surrogate consent.

You are being asked to serve as the Surrogate for \_\_\_\_\_\_\_, who is called the Subject in this document. You are being asked to give permission for the Subject to participate in this Study. Your decision should be based on the Subject's individual health care instructions and other wishes, if known, or on your best estimation of what you believe are the Subject's personal values and what the Subject would choose for himself/herself.

### Would the person for whom you are signing consent want to take part in this Study?

This form tells you about this Study. After reading this entire form and having this Study explained to you by someone conducting this Study, you can decide if you think the person for whom you are authorizing consent would want to take part in this Study. It is important to note that the person for whom you are signing consent does not have to take part in this Study in order to receive medical care outside this Study.

# What will happen if you, as the Surrogate, do not enroll the Subject in this Study, or if the Subject, or you as the Surrogate, later does not want the Subject to participate in this Study?

The Surrogate can decide not to enroll the Subject. The Subject or the Surrogate can decide to discontinue at any time the Subject's participation in this Study. Any decision by the Surrogate not to enroll the Subject or by the Subject or the Surrogate to discontinue the Subject's participation shall not affect the Subject including the Subject's receipt of medical care outside the Study. The Subject may withdraw without penalty and without loss of any benefits to which s/he are entitled.

Regardless of the Surrogate's consent, the Investigator can take the Subject out of this Study at any time because it would not be in the Subject's best interest to stay in it.

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

### SIGNATURE PAGE WHEN SUBJECT REQUIRES A SURROGATE (OR LAR)

### AGREEMENT TO PARTICIPATE

| 1. Surrogate Consent: The purpose and procedures for this Study have been described to me verbally and in writing. My questions about this Study have been answered and I have been provided with information about who to contact with additional questions. |
|---|
| As Surrogate, I freely give my consent to have |
| Signature of Surrogate Printed name of Surrogate Date |
| 2. Signature of Investigator/Individual Obtaining Consent: |
| To the best of my ability, I have explained and discussed the full contents of the study including all of the information contained in this consent form. All questions of the research subject and those of his/her parent or legally authorized representative have been accurately answered. |
| Investigator/Person Obtaining Consent (printed name): |
| Signature:Date: |
| 3. Signature of Consent Process Witness: |
| I have observed the consent process, which included a description of the purposes and procedures of this Study and an opportunity for questions and answers about this Study. I attest that I am not the subject, his/her guardian or authorized representative, or a researcher on this study and can attest that the requirements for informed consent to the medical research have been satisfied. |
| Signature of Witness Printed Name of Witness Date |

Feasibility and Safety Study

PI: Baburao Koneru, MD, MPH

## RUTGERS New Jersey Medical School

Department of Surgery/Division of Liver Transplant and Hepatobiliary Surgery Rutgers, The State University of New Jersey 185 South Orange Avenue, Medical Science Building G595 Newark, NJ 07103

p. 973-972-2408 f. 973-972-0006

### III. CONSENT TO TAKE PART IN A RESEARCH STUDY FOR INDIVIDUALS ENROLLED UNDER PRIOR SURROGATE CONSENT

**TITLE OF STUDY:** Remote Ischemic Conditioning (RIC) in Recipients of Brain Death Donor Livers – A Feasibility and Safety Study

### Principal Investigator: Baburao Koneru, MD, MPH

| Under certain circumstances, someone can give consent for another person to take part in a |
|---|
| research study. This person is providing "surrogate consent." The surrogate can make choices |
| for the subject, if the subject is not able to make choices for him or herself. In fact, since |
| you have been enrolled in this research study by your surrogate, |
| , you have occar and a second a second and a second a second and a second a second and a second a second and a second and a second a sec |

Now that you can make your own decision about whether or not to participate in this research study, please carefully review this entire form, **including both Section I and Section II**, which tells you about the research study. After reading through this form and having the research explained to you by someone conducting this research, you can decide if you wish to remain in the study or to withdraw. Your decision to withdraw will not affect the medical treatment you receive at the University.

Feasibility and Safety Study PI: Baburao Koneru, MD, MPH

### SIGNATURE PAGE WHEN SUBJECT WAS FORMERLY ENROLLED BY A SURROGATE (OR LAR)

| <b>DI</b> Modulo di la constanti di |
|---|
| AGREEMENT TO PARTICIPATE |
| 1. Subject Consent: |
| I have read this entire form, or it has been read to me, and I believe that I understand what has been discussed. All of my questions about this form or this study have been answered. |
| I agree OR I do not agree to continue to participate. |
| Subject Name: |
| Subject Signature:Date: |
| 2. Signature of Investigator/Individual Obtaining Consent: |
| To the best of my ability, I have explained and discussed the full contents of the study including all of the information contained in this consent form. All questions of the research subject have been accurately answered. |
| Investigator/Person Obtaining Consent: |
| Signature:Date: |
| 3. Signature of Consent Process Witness: |
| I have observed the consent process, which included a description of the purposes and procedures of this Study and an opportunity for questions and answers about this Study. I attest that I am not the subject, his/her guardian or authorized representative, or a researcher on this study and can attest that the requirements for informed consent to the medical research have been satisfied. |
| Signature of Witness Printed Name of Witness Date |